CLINICAL TRIAL: NCT03732040
Title: Miswak Versus Standard Measures to Prevent the Incidence of Caries Young Egyptian Adults: A Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Rashad Omar, Miswak versus standard measures to prevent the incidence of caries young Egyptian adults: A Randomized Controlled Clinical Trial, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4112018
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Toothbrushing; Fluorides

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standerd preventive measures (Sham Comparator): tooth brushing twice daily with fluoride tooth paste and dental flossing and mouthwash
  Interventions: Other: Standard preventive measures (tooth brushing , interdental cleaning and mouth rinse use containing CHX and Fluoride)
- miswak stick (Experimental): use of miswak stick twice daily
  Interventions: Other: miswak stick
- Use of Miswak plus tooth brushing and tooth paste (Experimental): use of miswak stick and tooth brush with fluoride toothpaste twice daily
  Interventions: Other: Miswak plus tooth brushing and tooth paste

INTERVENTIONS:
Other: miswak stick — miswak stick use as preventive hygiene measures
  Arms: miswak stick
Other: Miswak plus tooth brushing and tooth paste — use of miswak stick with tooth brushing and fluoride toothpaste for oral hygiene measures
  Arms: Use of Miswak plus tooth brushing and tooth paste
Other: Standard preventive measures (tooth brushing , interdental cleaning and mouth rinse use containing CHX and Fluoride) — use toothbrush with fluoride toothpaste and interdental cleaning by dental flossing and use mouth wash containing chlorohexadine
  Arms: standerd preventive measures

SUMMARY:
Objectives:

Aim of the study The objective is to conduct an RCT to evaluate the effectiveness of miswak in comparison with standard caries preventive measures for the prevention of new carious lesions in high caries risk patients.

-Research hypothesis (alternative hypothesis): This study will be designed to test the alternative hypothesis that using miswak in addition to standard preventive measures will show significant difference over using standard preventive measures alone in preventing incidence of new carious lesions in high caries risk patients.

DETAILED DESCRIPTION:
- General procedures The study will be announced at the Faculty of Oral and Dental Medicine, 6 October University campus to encourage interested students to participate in the study.

Interested participants will be screened at Conservative Department clinic for eligibility by (M.M). Eligible participants will be assessed using caries risk assessment tool by (R.R.).

Eligible participants will be randomly divided into three groups 1st group will follow only standard preventive measures(tooth brushing and tooth paste plus interdental cleaning and mouth rinse using CHX and Fluoride) , 2nd group will use miswak for oral hygiene measures and 3rd group will use of miswak plus tooth brushing and tooth paste.

Before starting the study the eligible participants will undergo supragingival, subgingival scaling and prophylaxis polishing, then any carious cavity, or defective restoration will be treated and filled with resin composite restoration.

New set of manual brushes and dental floss will be given to the participants, after they are properly trained for the correct brushing and flossing technique. The participants will be asked to brush their teeth twice a day with fluoride tooth paste and to clean their teeth interdentally with dental floss once a day every day till the end of the study(Group 1 and 3 only) 11b- Preparation of miswak

* Procedure of preparing Miswak:

Miswak has its own unique aspects that must be adapted prior to use for the best results. The functional end of a thin bark piece is striped off followed by chewing. Chewing of miswak separates fibers and giving it a brush like appearance that helps in cleaning the teeth easily. The recommended length for a stick is about 15 cm so that it can easily be grasped along with ease to carry around, whereas, the diameter is preferred to be <1 cm.(16) There are two methods documented to hold the miswak. One is the three finger grip technique and the other is five finger grip technique The aim of both techniques is to make sure that all surfaces of the teeth are accessible and cleaned with convenience and controlled movements of the stick in the oral cavity. In order to clean the tooth surfaces, the fibers of miswak should be held perpendicular to the tooth surface and gently moved in up and down motions, directed away from the gingival margins on both the buccal and lingual surfaces(17) .

11c-For the intervention group After recording the primary data, Miswak will be given to the intervention group and they will be trained and asked to use it two times per day. The demonstrations and instructions for chewing stick users will include the technique of preparation of working end of chewing sticks and its appropriate brushing technique. The sticks which are not prepared are instructed to be refrigerated. (13)(14).(group 2 and 3)

- For the control group Participants in this group will follow only the standard preventive measures which is brushing twice a day after breakfast and before bed time and daily flossing interdentally before bed time and mouth rinse containing CHX and fluoride.

In all study groups if any patient during the period of the study develops any carious cavity, the affected tooth will be treated immediately and restored with resin composite restoration.

. Outcomes: Visual inspection to detect presence or absence of new caries lesions will be done according to WHO guidelines by using CPI Probe (15).

ELIGIBILITY:
Inclusion Criteria:

* • patients with High caries risk

  * 18-25 years
  * Males or females
  * Medically free patients
  * Patients approving to participate in the study

Exclusion Criteria:

* Patients were on antibiotic therapy or corticosteroid therapy for 30 days before the examination
* Patients had history of professional cleaning in the last 15 days
* Patients with exposed pulp
* Evidence of parafunctional habits
* Patients with developmental dental anomalies
* Patients undergoing or will start orthodontic treatment
* Patients with removable prosthesis
* Periapical Abscess or Fistula

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of new caries lesions | 12 months
  visual tactil inspection

CONTACTS AND LOCATIONS:
Locations (1):
- 6Th of October University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided